CLINICAL TRIAL: NCT03194035
Title: Per Effort Study of Inflammatory Consequences of an Ultra Endurance Race (165km)
Brief Title: Inflammation in an Ultra Endurance Race
Acronym: TRAIL-INFLA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, Principal Investigator, Hôpital Necker-Enfants Malades
Other Study IDs: TRAIL-INFLA
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Inflammation; Inflammatory Response
Keywords: inflammation; exercise; ultra endurance
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sample — Study per and post-exertional changes in proinflammatory biological (IL1, IL6, TNF alpha, HMG beta1 and CRP) and anti inflammatory parameters (IL4, IL10 and IL13, TGF beta, LPS, lipoproteins, lipids) during an ultra endurance race.

SUMMARY:
The aim of this study is to study the per and post-exertional variations of the pro and anti inflammatory markers during an ultra-endurance race in healthy volunteers.

DETAILED DESCRIPTION:
Study per and post-exertional changes in proinflammatory biological (IL1, IL6, TNF alpha, HMG beta1 and CRP) and anti inflammatory parameters (IL4, IL10 and IL13, TGF beta, LPS, lipoproteins, lipids) during an ultra endurance race.

ELIGIBILITY:
Inclusion Criteria:

1. Male older than 18 years,
2. Completion of an ultra-endurance race (distance greater than 50 kilometers) during the 24 months preceding the race.
3. Affiliation or beneficiary of a social security.

Exclusion Criteria:

1. Age lower than 18 years,
2. Subjects with a medical history (pulmonary pathology, cardiac, hypertension) or with a significant chronic inflammatory disease observed during the inclusion visit (the day before the race).
3. Female.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 healthy adult volunteers amateurly participating in the "100 miles South of France 2017 race ©" recruited electronically using an announcement on the race website.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-17 (Estimated)

PRIMARY OUTCOMES:
Per and post-exertional variations of IL1 during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of IL1 blood level
Per and post-exertional variations of IL6 during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of IL6 blood level
Per and post-exertional variations of TNF alpha during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of TNF alpha blood level
Per and post-exertional variations of HMG beta during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of HMG beta blood level
Per and post-exertional variations of CRP during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of CRP blood level
Per and post-exertional variations of IL4 during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of IL4 blood level
Per and post-exertional variations of IL10 during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of IL10 blood level
Per and post-exertional variations of IL13 during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of IL13 blood level
Per and post-exertional variations of lipids during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of lipids blood level
Per and post-exertional variations of LPS during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of LPS blood level
Per and post-exertional variations of lipoprotein during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of lipoprotein blood level
Per and post-exertional variations of TGF beta during an ultra-endurance race in healthy volunteers. | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  In this study, the investigators will measure variations of TGF beta blood level

IPD SHARING:
Plan to Share IPD: No